CLINICAL TRIAL: NCT03866408
Title: Insulin Regulation of Lipolysis and Lipolysis Proteins
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17-009837; 2R01DK040484-30 (NIH)
Record Dates: First submitted 2018-12-13; First posted 2019-03-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: adipose tissue
MeSH Terms: conditions — Obesity | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: immediate weight loss (placebo) will be compared with deferred weight loss (placebo) to determine the effects of weight loss alone immediate weight loss placebo will be compared with deferred weight loss pioglitazone to determine the effects of weight loss vs. pioglitazone deferred weight loss placebo will be compared with deferred weight loss pioglitazone to determine the effects of pioglitazone alone deferred weight loss placebo will be compared with deferred weight loss pioglitazone to determine the effects of weight loss alone vs. previous exposure to pioglitazone immediate weight loss placebo and deferred weight loss placebo will be pooled to create a larger group to determine the effects of weight loss on outcome variables
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Immediate weight loss - placebo (Active Comparator): Upper body obese participants randomized to this group; all will begin their immediate participation in a comprehensive lifestyle obesity treatment program after completion of baseline studies. Half of the volunteers will be randomized to placebo during this period.
  Interventions: Behavioral: Immediate weight loss; Drug: Placebo
- Deferred control group - placebo (Placebo Comparator): After baseline studies, UBO participants randomized to this group will wait without any intervention for 4 months, with continued monitoring to assure weight stability - this group will be the half of volunteers randomized to deferred weight loss intervention that are also randomized to placebo. At the end of this 'wait' period they will be enrolled in the same comprehensive lifestyle obesity treatment program for 4 months, but without placebo.
  Interventions: Behavioral: Deferred weight loss; Drug: Placebo
- Immediate weight loss - pioglitazone (Active Comparator): Upper body obese participants randomized to this group; all will begin their immediate participation in a comprehensive lifestyle obesity treatment program after completion of baseline studies. Half of the volunteers will be randomized to pioglitazone during this period.
  Interventions: Behavioral: Immediate weight loss; Drug: Pioglitazone
- Deferred group - pioglitazone (Active Comparator): After baseline studies, UBO participants randomized to this group will wait without any intervention for 4 months, with continued monitoring to assure weight stability - this group will be the half of volunteers randomized to deferred weight loss intervention that are randomized to pioglitazone. They will be monitored to prevent the usual but modest weight gain associated with pioglitazone. They will be on pioglitazone during the 'wait' period.
  At the end of this 'wait' period they will be enrolled in the same comprehensive lifestyle obesity treatment program for 4 months, but without pioglitazone.
  Interventions: Drug: Pioglitazone; Behavioral: Deferred weight loss

INTERVENTIONS:
Behavioral: Immediate weight loss — Upper body obese subjects will undergo behavioral intervention with a life coach and a physical activity program of their choice for 4 months.
  Arms: Immediate weight loss - pioglitazone; Immediate weight loss - placebo
Drug: Pioglitazone — Upper body obese subjects will be block randomized to pioglitazone or placebo at enrollment.
  Arms: Deferred group - pioglitazone; Immediate weight loss - pioglitazone
Behavioral: Deferred weight loss — Upper body obese subjects will complete a weight-stable period of 4 months and subsequently undergo behavioral intervention with a life coach and a physical activity program of their choice for 4 months.
  Arms: Deferred control group - placebo; Deferred group - pioglitazone
Drug: Placebo — Upper body obese subjects will be block randomized to pioglitazone or placebo at enrollment.
  Arms: Deferred control group - placebo; Immediate weight loss - placebo

SUMMARY:
These studies will define the abnormalities in the adipocyte proteins that are involved in the failure of insulin to suppress lipolysis normally in humans with upper body obesity and will help discover the mechanism by which pioglitazone, a medication used to treat type 2 diabetes and improve insulin resistance, improves insulin-regulation of adipocyte fatty acid metabolism.

DETAILED DESCRIPTION:
1. The investigators will determine whether impaired insulin-induced suppression of lipolysis (as measured by IC50) is related to the above mentioned lipolysis proteins in groups of volunteers known to vary widely with regards to abdominal adipocyte size and regulation of adipose tissue lipolysis.
2. The investigators will determine whether the improved insulin regulation of lipolysis resulting from treatment with the PPARγ agonist pioglitazone, with or without weight loss, can be linked to specific changes in sets of PPARγ-responsive adipocyte lipolysis proteins in UBO adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between the ages of 18 and 55.
* Women will be premenopausal
* Non obese adults BMI between 18-25
* Obese BMI 30-38

Exclusion Criteria, Pioglitazone package insert of contraindications for use:

* Initiation in patients with established New York Heart Associations (NYHA) class III or IV Heart failure.
* Use in patients with known hypersensitivity to pioglitazone or any other component of ACTOSE.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adipocyte response to insulin - perilipin 1 and FSP27 relative to HSL and ATGL | 4-9 months
  In response to weight maintenance vs. weight loss with pioglitazone vs. placebo, insulin regulation of lipolysis in upper body obese as measured by insulin IC50 for palmitate flux and compared to adipocyte perilipin 1 and FSP27 relative to HSL and ATGL.
Adipocyte response to insulin - adipocyte G0S2 relative to ATGL. | 4-9 months
  In response to weight maintenance vs. weight loss with pioglitazone vs. placebo, insulin regulation of lipolysis in upper body obese as measured by insulin IC50 for palmitate flux and compared to adipocyte G0S2 relative to ATGL.
Adipocyte response to insulin - adipocyte CGI-58 relative to ATGL | 4-9 months
  In response to weight maintenance vs. weight loss with pioglitazone vs. placebo, insulin regulation of lipolysis in upper body obese as measured by insulin IC50 for palmitate flux and compared to adipocyte CGI-58 relative to ATGL.
Adipocyte response to insulin - perilipin 1, ATGL and HSL phosphorylation | 4-9 months
  In response to weight maintenance vs. weight loss with pioglitazone vs. placebo, insulin regulation of lipolysis in upper body obese as measured by insulin IC50 for palmitate flux and compared to adipocyte perilipin 1, ATGL and HSL phosphorylation in response to insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials